CLINICAL TRIAL: NCT06438913
Title: The Improvement of Cough Outcomes After Tezepelumab Treatment in Korean Severe Asthma Patients With Airway Hyperresponsiveness
Brief Title: Tezepelumab Treatment in Korean Severe Asthma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Bum Kim, Principal Investigator, Asan Medical Center
Other Study IDs: 2024-0215
Record Dates: First submitted 2024-05-17; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Tezepelumab — Tezepelumab blocks thymic stromal lymphopoietin (TSLP), an epithelial cytokine suggested to be important in the initiation and continuation of airway inflammation.

SUMMARY:
There is no study that systematically evaluated the effect of Tezepelumab on cough, and based on this background, the present researchers aimed to evaluate the effect of Tezepelumab treatment in patients with severe asthma who complain of cough using the Leicester Cough Questionnaire, a cough-related quality of life measurement tool.

ELIGIBILITY:
Inclusion Criteria:

1. Severe asthma patients aged 19 or older and 79 or younger
2. Cases diagnosed as asthma by an expert and classified as severe asthma according to the 2014 ATS/ERS guidelines

   - Patients who require the use of high-dose inhaled steroids and additional control agents or systemic steroids for more than 50% of the year to control symptoms. Or, if asthma is not controlled even with the medication. Here, uncontrolled asthma means that any one of the following is satisfied.
   1. ACT score less than 20 or 'not well controlled' according to GINA guideline
   2. frequent exacerbations; Requires systemic steroid administration (over 3 consecutive days) more than twice in the previous year If you did
   3. severe exacerbation; A condition that required hospitalization, admission to an intensive care unit, or application of a ventilator in the previous year If you have been angry at least once
   4. airflow restrictions; FEV1 < 80%
3. If a cough is due to asthma according to a doctor and the cough onset scale (cough visual analogue scale, cough VAS) satisfies 30 or more points out of 100.
4. If a positive result is confirmed in the methacholine (or mannitol) bronchial challenge test (if the bronchial challenge test result is not available or the test is difficult to proceed, it can be replaced with a positive bronchodilator response test)

Exclusion Criteria:

1. Minors under 19 years of age, senior citizens over 79 years of age
2. If there is a history of use of other biological agents within 3 months prior to study registration
3. Cases where there was an acute exacerbation requiring a steroid burst (total 90mg prednisolone or more) during the 4-week screening period before study registration (possible for long-term prednisolone users)
4. Cases accompanied by clinically serious respiratory disease in addition to severe asthma
5. When accompanied by hypereosinophilic syndrome, ABPA, EGPA
6. When it is difficult to evaluate asthma alone due to severe respiratory disease
7. Pregnant women

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-12 (Estimated); Primary Completion 2025-05-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Effects of Tezepeluma on Cough | 1years
  The effectiveness of Tezepelumab on cough was assessed by comparing the LCQ score at 1 and 12 months of administration with the LCQ score at the time of registration.